CLINICAL TRIAL: NCT03176316
Title: The Use of Oral Naloxone to Prevent Post Spinal Fusion Ileus
Acronym: FusionIleus
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated by the Institutional Review Board.
Sponsor: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 209439
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Ileus; Fusion of Spine
Keywords: ileus; fusion of spine
MeSH Terms: conditions — Ileus | interventions — Naloxone

STUDY DESIGN:
Intervention Model Description: All participants who agree to participate in the study and meet the inclusion and exclusion criteria may receive the planned study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Naloxone (Experimental): 1 mg/ml oral solution administered enterally every eight hours for 48 hours
  Interventions: Drug: Naloxone

INTERVENTIONS:
Drug: Naloxone — Naloxone is an opioid antagonist (i.e., a medication used to reverse or reduce the effects of opioids)

SUMMARY:
Postoperative ileus and opioid induced constipation are well-known post-operative complications. Previously, research has shown that using peripherally acting opioid antagonists can help alleviate the condition. There has not been a prospective study to investigate whether use of peripherally acting opioid antagonists are effective in preventing post-operative ileus in patients having spinal fusion surgeries.

DETAILED DESCRIPTION:
Post operative ileus is a well-known complication following spinal fusion surgery. There has been some literature to demonstrate the safety and efficacy of oral naloxone to decrease the time to bowel movements after gastrointestinal surgery, to date, there have been no studies within the spine fusion literature to investigate oral naloxone's effects on the time to bowel movements.

The aim of the present study is to use the previously established protocols and doses established in the gastrointestinal literature to see whether oral naloxone can decrease the time to first bowel movements.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they are having an in-patient spinal fusion procedure, are 18 years or older, post and post-operative pain control plan includes opioid medications.

Exclusion Criteria:

* Pregnancy, age < 18, nursing, or documented allergy to naloxone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Nockels, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data with other researchers

REFERENCES:
- [Background] Arpino PA, Thompson BT. Safety of enteral naloxone for the reversal of opiate-induced constipation in the intensive care unit. J Clin Pharm Ther. 2009 Apr;34(2):171-5. doi: 10.1111/j.1365-2710.2008.00982.x. PMID 19250137
- [Background] McNicol E, Boyce DB, Schumann R, Carr D. Efficacy and safety of mu-opioid antagonists in the treatment of opioid-induced bowel dysfunction: systematic review and meta-analysis of randomized controlled trials. Pain Med. 2008 Sep;9(6):634-59. doi: 10.1111/j.1526-4637.2007.00335.x. PMID 18828197
- [Background] Fineberg SJ, Nandyala SV, Kurd MF, Marquez-Lara A, Noureldin M, Sankaranarayanan S, Patel AA, Oglesby M, Singh K. Incidence and risk factors for postoperative ileus following anterior, posterior, and circumferential lumbar fusion. Spine J. 2014 Aug 1;14(8):1680-5. doi: 10.1016/j.spinee.2013.10.015. Epub 2013 Oct 31. PMID 24184650
- [Background] Meissner W, Leyendecker P, Mueller-Lissner S, Nadstawek J, Hopp M, Ruckes C, Wirz S, Fleischer W, Reimer K. A randomised controlled trial with prolonged-release oral oxycodone and naloxone to prevent and reverse opioid-induced constipation. Eur J Pain. 2009 Jan;13(1):56-64. doi: 10.1016/j.ejpain.2008.06.012. Epub 2008 Aug 31. PMID 18762438
- [Background] Meissner W, Schmidt U, Hartmann M, Kath R, Reinhart K. Oral naloxone reverses opioid-associated constipation. Pain. 2000 Jan;84(1):105-109. doi: 10.1016/S0304-3959(99)00185-2. PMID 10601678
- [Background] Sykes NP. An investigation of the ability of oral naloxone to correct opioid-related constipation in patients with advanced cancer. Palliat Med. 1996 Apr;10(2):135-44. doi: 10.1177/026921639601000208. PMID 8800821
- [Background] Lee J, Shim JY, Choi JH, Kim ES, Kwon OK, Moon DE, Choi JH, Bishop MJ. Epidural naloxone reduces intestinal hypomotility but not analgesia of epidural morphine. Can J Anaesth. 2001 Jan;48(1):54-8. doi: 10.1007/BF03019815. PMID 11212050

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on September 20, 2017 and ended on February 20, 2020 when the Institutional Review Board placed the project on administrative hold. Recruitment occurred at a Loyola University Medical Center clinic.
Groups:
- Naloxone: Naloxone is an opioid antagonist (i.e., a medication used to reverse or reduce the effects of opioids). The study administers 1 mg/ml oral solution enterally every eight hours for 48 hours.
Period: Overall Study
Arm/Group | Naloxone
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Naloxone
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Information on participant age was only collected for 23 participants.
  years
    number analyzed (Participants) | 23
    (all) | 65.91 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 31
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Time to First Bowel Movement
Description: We will monitor the patients' bowel movements and record the time to the first bowel movement in hours
Time Frame: 1 week
Population: The research team collected outcome data on one participant. The Institutional Review Board terminated the study early due to non-compliance with continuing review requirements.
Measure: Number; unit: Hours
Arm/Group | Naloxone
Number analyzed (Participants) | 1
Hours | 43.62

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 years and 5 months
Arm/Group | Naloxone
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03176316/Prot_SAP_000.pdf